CLINICAL TRIAL: NCT01849276
Title: A Phase I Study of Metformin and Cytarabine for the Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Metformin+Cytarabine for the Treatment of Relapsed/Refractory AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jessica Altman, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 11H03; NCI-2011-01084 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00048047 (Other: Northwestern University IRB#)
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Blastic Phase Chronic Myelogenous Leukemia; Recurrent Adult Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Blast Crisis | interventions — Metformin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor and chemotherapy) (Experimental): Patients receive metformin hydrochloride orally twice a day on days 1-15 and cytarabine IV over 3 hours twice on days 4-10.
  Interventions: Drug: metformin hydrochloride; Drug: cytarabine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: metformin hydrochloride — Given orally
  Other Names: Glucophage
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The purpose of the study is to determine if metformin in combination with cytarabine is safe and effective. Participants in this research study have acute myeloid leukemia (AML) that has come back after initial treatment or has not gone away with initial therapy.There is evidence that metformin directly kills leukemia cells. Laboratory data have also shown that combinations of metformin with cytarabine are more efficient than each agent alone in killing leukemia cells in the laboratory.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of metformin (metformin hydrochloride) in combination with cytarabine in relapsed/refractory AML.

II. Define the dose limiting toxicity (DLT) of metformin in combination with cytarabine in relapsed/refractory AML.

SECONDARY OBJECTIVES:

I. Remission rate. II. Overall survival (OS). III. Disease-free survival (DFS). IV. Length of remission.

OUTLINE: This is a dose-escalation study of metformin hydrochloride in combination with Cytarabine.

Patients receive metformin hydrochloride orally (PO) twice daily (BID) on days 1-15 and cytarabine intravenously (IV) over 3 hours BID on days 4-10.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory disease must have morphologic proof (from bone marrow aspirate, smears or touch preps of bone marrow biopsy) of AML with >= 10% blasts within two weeks (14 days) prior to initiation of therapy

  * All immunophenotype and cytogenetic/molecular groups are eligible for participation except for acute promyelocytic leukemia (APL) (as proven by the presence of promyelocytic leukemia/retinoic acid receptor alpha [PML-RARα])
* Patients must demonstrate one of the following:

  * Relapse after first complete remission
  * Refractory to conventional induction chemotherapy (failure to respond to 1 or more cycles of daunorubicin and cytarabine) or to re-induction
* Patients with previously untreated AML are candidates if they are unable to receive anthracyclines, and have documented AML with >= 20% blasts within one week prior to enrollment
* Patients with chronic myelogenous leukemia (CML) in myeloid blast crisis are eligible if their disease has failed to respond, and/or they are intolerant, to the available tyrosine kinase inhibitors (TKIs)
* Serum total and direct bilirubin =< upper limit of normal (ULN)
* Serum creatinine < 1.4 mg/dl in females and < 1.5 mg/dl in males, and creatinine clearance > 60 mL/min
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST])/serum glutamic pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< ULN
* Bicarbonate within the normal range of the hospital lab (24-32 mmol/L)
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Females of childbearing potential and sexually active males must agree to use an accepted and effective method of contraception while on study
* Childbearing potential is defined as any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has NOT undergone a hysterectomy or bilateral oophorectomy; OR
  * Has NOT been naturally postmenopausal for at least 12 consecutive months (i.e. has had menses at any time in the preceding 12 consecutive months)
* Patients with a history of central nervous system (CNS) leukemia are eligible if they are not symptomatic from current CNS involvement

  * If there is CNS involvement that is known prior to enrollment or identified subsequently, it will be treated accordingly
* Patients may have received therapy for other malignancies, as long as they have completed therapy at least 6 months prior to study entry and be deemed to have a life expectancy of at least 2 years with regard to that malignancy
* All patients must have given signed, informed consent prior to registration on study

Exclusion Criteria:

* Patients who have received chemotherapy or radiotherapy within 4 weeks prior to enrollment are NOT eligible for participation

  * The exception to this is patients who are refractory to conventional initial induction chemotherapy (=< 2 courses) or to first radiation (1 course); patients must have morphologic proof (from bone marrow aspirate, smears, or touch preps of marrow biopsy) of AML with > 10% blasts within 2 weeks prior to initiation of study therapy; the last dose of cytotoxic therapy (NOT including hydrea, which is allowed) must have been given >= 14 days prior to initiation of study therapy
* Patients with a history of diabetes mellitus (DM) treated with metformin are NOT eligible for participation
* Patients who are pregnant or breast feeding are NOT eligible for participation due to the lack of knowledge regarding the effects of the drugs on the fetus and during breast feeding
* Patients with any intercurrent organ damage or medical problems that would prohibit therapy are NOT eligible for participation
* Patients with any active, uncontrolled infection are NOT eligible for participation
* Patients who are receiving therapy for another active malignancy are NOT eligible for participation

  * The exception to this is squamous cell carcinoma or basal cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2016-01-21 (Actual); Study Completion 2016-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Altman, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual July 29, 2013 with an accrual goal of between 19 to 28 participants in a 3 + 3 dose escalation design to find the maximum tolerated dose of metformin in combination with cytarabine. The study was closed permanently on January 21 2016 due to slow accrual.
Period: Registered to the Study
Arm/Group | Treatment (Enzyme Inhibitor and Chemotherapy)
Started | 2
Completed | 2
Not Completed | 0
Period: Completed Treatment
Arm/Group | Treatment (Enzyme Inhibitor and Chemotherapy)
Started | 2
Completed | 2
Not Completed | 0
Period: Followed for Survival for 5 Years
Arm/Group | Treatment (Enzyme Inhibitor and Chemotherapy)
Started | 2
Completed | 0
Not Completed | 2
Not completed — Death | 1
Not completed — Early termination of the study | 1

BASELINE CHARACTERISTICS:
Population: Two participants were enrolled and treated on the study before the study closed due to slow accrual
Arm/Group | Treatment (Enzyme Inhibitor and Chemotherapy)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Toxicity by Assessing the Adverse Events of Metformin and Cytarabine
Description: To determine the maximum tolerated dose (MTD) by assessing the adverse events of metformin in combination with cytarabine in evaluating toxicity. Assessments will occur daily during cytarabine administration and at least twice weekly following treatment until blood count recovery.
Time Frame: Checked daily during administration of cytarabine and at least 2x weekly following therapy until desired blood counts acheived (maximum 15 days)
Population: Adverse events that were assessed to be either possibly or unlikely related to treatment on study (i.e. relationship between treatment and adverse event could not be ruled out)
Measure: Number; unit: Adverse events related to treatment
Arm/Group | Treatment (Enzyme Inhibitor and Chemotherapy)
Number analyzed (Participants) | 2
Adverse events related to treatment
  Grade 1 | 4
  Grade 2 | 6
  Grade 3 | 2
  Grade 4 | 0

2. Primary Outcome: Study Treatment Dose Toxicity Will be Evaluated by Measurement of Adverse Events Experienced While on Treatment
Description: Determination of Dose Limiting Toxicity (DLT) as evidenced by adverse events due to toxicity from study treatment. If no DLT is observed, then 3 patients will be enrolled in the next dose escalated cohort. If one DLT is seen in the first 3 patients, then an additional 3 patients will be enrolled at the same dose cohort. If 0-1 in 6 patients experience a DLT this dose will be considered tolerable and the next dose escalated cohort with enroll 3 patients. If 2 or more in 6 patients experience a DLT, the maximum tolerated dose (MTD) will have been exceeded and the next cohort will enroll 3 patients at a reduced dose.
Time Frame: as for outcome 1
Population: The study was terminated early due to slow accrual, thus insufficient data was collected to be analysed.
Arm/Group | Treatment (Enzyme Inhibitor and Chemotherapy)
Number analyzed (Participants) | 0

3. Secondary Outcome: Remission Rate
Description: Patients will be evaluated for remission status in response to therapy.
Time Frame: Every 3 months for 2 years, and then every 6 months for 5 years post-treatment
Population: The study was terminated early due to slow accrual. As a result no data was collected or analyzed for this outcome measure.
Arm/Group | Treatment (Enzyme Inhibitor and Chemotherapy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Description: Patients will be followed-up with from the initiation of study treatment until progression of disease or for up to 5 years, whichever comes first.
Time Frame: Every 3 months for 2 years, and then every 6 months for 5 years post-treatment
Population: as for outcome 3
Arm/Group | Treatment (Enzyme Inhibitor and Chemotherapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Disease-free Survival
Description: Evaluation of Disease-Free Survival will defined as the time from the initiation of study treatment until the time of disease relapse.
Time Frame: Every 3 months for 2 years, and then every 6 months for 5 years post-treatment
Population: as for outcome 3
Arm/Group | Treatment (Enzyme Inhibitor and Chemotherapy)
Number analyzed (Participants) | 0

6. Secondary Outcome: Length of Remission
Description: Patients will be followed-up with to determine Remission length which is defined as the time from attainment of remission to relapse of disease.
Time Frame: From date of remission of disease to date of relapse (maximum of 5 year follow-up)
Population: as for outcome 3
Arm/Group | Treatment (Enzyme Inhibitor and Chemotherapy)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Bone Marrow and Blood Samples Will be Taken Prior to Study Treatment to Determine Number of Leukemic Progenitor Cells
Time Frame: At baseline prior to study treatment
Population: as for outcome 3
Arm/Group | Treatment (Enzyme Inhibitor and Chemotherapy)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Immunoblotting
Description: Bone marrow and/or blood samples taken prior to initiation of treatment will be used in Immunoblotting studies to observe enzyme and protein activity.
Time Frame: At baseline prior to study treatment
Population: as for outcome 3
Arm/Group | Treatment (Enzyme Inhibitor and Chemotherapy)
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Identical Immunoblotting
Description: Identical immunoblotting studies may also be performed using blood samples taken prior to start of treatment.
Time Frame: At baseline prior to study treatment
Population: as for outcome 3
Arm/Group | Treatment (Enzyme Inhibitor and Chemotherapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collect cover a 7 month period before the study was terminated early due to slow accrual
Arm/Group | Treatment (Enzyme Inhibitor and Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor and Chemotherapy) (N=2)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Other-Transminitis (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor and Chemotherapy) (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Elevated D-Dimer (Blood and lymphatic system disorders) | 1 (1)
Elevated INR (Blood and lymphatic system disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage - Hematochezia (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (5)
Pleural infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (3)
White blood cell decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminema (Metabolism and nutrition disorders) | 1 (7)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Symptomatic Bartholin gland (Reproductive system and breast disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study terminated early due to slow accrual and there was not sufficient data collected for statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes